CLINICAL TRIAL: NCT07311499
Title: A Study on Improving Sleep Quality in COPD Patients Through Inhalation Management Education by Nurses Using Video Conferencing Tools.
Brief Title: Improvement of Sleep in COPD Patients Through Inhalation Management Education by Nurse.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kumamoto University (Other)
Collaborators: Hiroshima University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: No. 2591; 24K14058 (Other Grant/Funding Number: Japan Society for the Promotion of Science); 202430036 (Other Grant/Funding Number: The Mitsubishi Foundation); Diversity initiatives (Other Grant/Funding Number: Kumamoto University)
Record Dates: First submitted 2025-09-08; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Lung Disease
Keywords: COPD; inhalation management education; sleep quality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- education intervention group (Active Comparator)
  Interventions: Behavioral: inhalation management education
- Normal care group (No Intervention): Provide a pamphlet tailored to the patient's inhalation device.

INTERVENTIONS:
Behavioral: inhalation management education — * During interviews with researchers, undergo a technical check. Then, practice inhalation techniques.
  * During interviews with researchers, discuss solutions to symptoms and problems encountered in daily life.
  * Participants implement the solutions decided upon during the observation period.
  * During the second intervention, assess whether the solutions were effective and, if not, consider alternative solutions.
  Arms: education intervention group

SUMMARY:
This study aims to investigate whether inhalation management education provided by nurses improves sleep quality in patients with COPD. Inhalation management education includes training in inhalation techniques and guidance on how to use medications when symptoms occur.

The main research question is:

・Does inhalation management education improve sleep quality in patients with COPD?

Researchers will determine whether inhalation management education improves sleep quality compared to no education.

Participants will:

* Participate in two interviews with researchers using video conferencing tools.
* Keep a diary recording their symptoms, sleep duration, and the frequency of rescue inhaler use.

DETAILED DESCRIPTION:
●Research participants, eligibility criteria, and exclusion criteria The study will include stable COPD patients who are outpatients at Kumamoto University Hospital, Kounan Hospital, or Iwakuni City Nishiki Central Hospital, which specialize in internal and respiratory medicine. Eligible participants must meet all of the following criteria and must not meet any exclusion criteria.

【Eligibility Criteria】

1. Aged 20 years or older at the time of informed consent.
2. Prescribed inhaled medications and have used them continuously for at least one month.
3. No prior experience with inhalation therapy required.
4. No hospitalization for COPD exacerbation within one month prior to study enrollment.
5. Patients with obstructive sleep apnea (OSAS) overlap syndrome (OVS) receiving nasal continuous positive airway pressure (CPAP) therapy are eligible if their symptoms are stable, as determined by a physician after CPAP initiation.
6. Able to operate a device such as an Android tablet, iPad, or computer; if not, participation is still acceptable if a caregiver can operate the device.
7. Individuals deemed to be in a stable condition by a physician and who have obtained permission.

【exclusion criterias】

1. Presence of other respiratory diseases such as asthma or interstitial pneumonia.
2. Presence of advanced cancer, including lung cancer.
3. Restricted chest movement due to chest deformity or trauma
4. Sleep-disordered breathing with a central apnea-hypopnea index (AHI) exceeding 50%.
5. Sleep-disordered breathing with a central AHI of more than half
6. Diagnosis of dementia or other psychiatric disorders.

   * Registration of study subjects The attending physician at the collaborating research institution will refer patients who meet the eligibility criteria for the study, and the principal investigator or research collaborator will obtain the patient's consent directly. The purpose and significance of the study, the methods, and ethical considerations will be explained verbally and in writing, and written consent will be obtained. After obtaining consent, a study subject identification code will be assigned, and the study subject will be registered in this study.
   * Allocation method A stratified block allocation will be performed using gender (male, female) and severity classification (GOLD Grade 1, 2, 3, 4) as allocation factors. The allocation of study participants to each treatment group will be conducted by Makiko Yamamoto at the Department of Basic Nursing Science, Kumamoto University Graduate School of Nursing.

   Following the pre-established random allocation table, participants will be sequentially assigned to each treatment group in the order of case registration, and a registration confirmation form will be issued, indicating the participant's registration number and treatment group. The allocation table will be retained by the allocation officer and will not be disclosed to the principal investigator or co-investigators.

   ●Sample size Target number of participants (Total: 34 cases) Intervention group: 17 cases Control group: 17 cases Number of participants expected to enroll(Total: 60 cases) Intervention group: 30 cases Control group: 30 cases There are no previous studies measuring the effect of inhalation management education on sleep quality. In previous studies, the average PSQI score for COPD patients was 8.3-11.5 points, and the PSQI cutoff value is 5.5 points. Assuming a change of 5.0 points in the average PSQI-J score after 3 months in the intervention group, the sample size required to maintain a two-sided test (significance level 5%) with 80% power is 17 cases per group. Considering that many participants are elderly and may have difficulty continuing to use computers or video conferencing tools, a higher dropout rate than usual is anticipated. Therefore, 30 participants per group, totaling 60 participants, will be enrolled in the study.

   ●Criteria for exclusion from analysis The definition of the analysis population is as follows.

   -Full Analysis Set (FAS) The FAS consists of all study subjects who provided informed consent, excluding the following study subjects.
   * Cases that do not meet the primary eligibility criteria (e.g., diagnosed with a disease outside the scope of the study, or found to have violated objectively determinable selection or exclusion criteria) • Cases with no post-randomization measurements -The population compliant with the study protocol (Per Protocol Set: PPS)

   The PPS is defined as the FAS excluding the following subjects:

   • Cases with unavailable measurements of the primary endpoint

   • Cases with major protocol violations (e.g., allocation errors, failure to meet eligibility criteria, non-compliance with medication)

   This study will clearly identify the breakdown of cancellations and dropouts by compiling data on the number of registered subjects who were excluded from the analysis population and the reasons for their exclusion, broken down by analysis population.

   ●Analysis and statistical methods for verifying evaluation items Statistical analysis will be performed using JMP Pro 18, with a significance level set at 5%.

   -Analysis of primary endpoints Primary endpoint: Change in PSQI-J at 3 months before and after the educational intervention The primary endpoint will be analyzed using the FAS. The change in PSQI-J scores will be calculated for each group, and independent t-tests will be performed to compare groups at a significance level (two-sided) of 5%. A similar analysis will be conducted using PPS as the analysis population as a secondary analysis.

   -Using FAS as the analysis population, the difference in the mean change in JESS, Japanese CAT, and HADS scores between groups will be analyzed using a paired t-test at a significance level of 5%. Similar analyses will also be conducted using PPS as the analysis population.

   In this study, baseline data for the primary outcome measure, PSQI, were missing at study registration. If PSQI-J was measured within one month of baseline (prior to the first intervention), that data was used to impute baseline data for PSQI-J. This method of data imputation may result in the presence of data from different measurement time points at baseline.

   However, since the PSQI-J reflects sleep quality over the past month and no interventions were conducted during that period, this method of data supplementation is considered appropriate. For other items, missing values will not be supplemented.

   Information on patients obtained at baseline from participants who withdrew from the study or withdrew their consent will be used for analysis if consent is obtained from the participants themselves, as it constitutes valuable data on inhalation techniques, inhalation education, and methods for current COPD patients.

   ●Criteria for discontinuing participation in research The principal investigator or co-investigator shall terminate the study if they determine that it is impossible to continue the study for any of the following reasons.

   <Termination Criteria>

   • If a research subject withdraws from the study or revokes their consent

   • If it is determined after registration that the subject no longer meets the eligibility criteria (inclusion/exclusion criteria)
   * If the subject requires emergency hospitalization and treatment due to worsening of the underlying disease
   * If the study cannot be continued due to worsening of complications
   * If the study cannot be continued due to adverse events
   * If the study is terminated
   * If the physician determines that termination of the study is appropriate for other reasons

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 20 years or older at the time of consent.
* Individuals who have been prescribed inhaled medications and have been using them continuously for more than one month.
* Prior experience with inhalation instruction is not required.
* Individuals who have not been hospitalized within one month prior to study participation due to exacerbation of COPD.
* Individuals with obstructive sleep apnea syndrome (OSAS) who are receiving treatment with continuous positive airway pressure (CPAP) therapy are eligible, provided that the physician determines that symptoms are stable following CPAP initiation.
* Participants must be able to operate devices such as Android, iPad, or computer. However, if a caregiver can operate the device, the participant's inability to do so is acceptable.
* Participants must be in a stable condition as determined by a physician and have obtained permission to participate.

Exclusion Criteria:

* Suffering from other respiratory diseases such as asthma or interstitial pneumonia
* Suffering from advanced cancer, including lung cancer
* Restricted chest movement due to chest deformity or trauma
* Suffering from diseases that cause respiratory distress, such as heart disease
* Suffering from sleep-disordered breathing with a central AHI of more than 50%
* Diagnosed with dementia or mental illness

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
The Japanese version of the Pittsburgh Sleep Quality Index： PSQI-J | Baseline, 2months and 3months
  The PSQI-J is a questionnaire that asks about sleep patterns over the past month. It consists of 19 self-reported items and seven factors: sleep quality, sleep onset time, sleep duration, sleep efficiency, sleep difficulty, use of sleep medication, and daytime sleepiness. A total score of 0 to 3 points (0 to 21 points) is calculated, and the higher the score, the more severe the sleep disorder is considered to be.

SECONDARY OUTCOMES:
Japanese Version of Epworth Sleepiness Scale：JESS | B0aseline, 2months and 3months
  This is a self-assessment of the degree of sleepiness in eight daily-life situations. Each item is scored from 0 to 3(0-24 points), with higher total scores indicating greater daytime sleepiness. If the total score is 11 or higher, it is likely that the patient has SAS (sleep apnea syndrome).
Apnea-Hypopnea Index | Baseline and 3 months
  Apnea-Hypopnea Index(AHI) is an index used to evaluate sleep apnea syndrome (SAS). It is calculated as the total number of observed apneas and hypopneas during sleep divided by the total sleep time (typically per hour). Diagnose with sleep apnea syndrome based on AHI>5.
Depth of REM sleep | Baseline and 3months
  During REM sleep, estimates include the number and duration of wakefulness episodes and the proportion of REM time spent awake. The more times it occurs, the more it is considered to be disrupting sleep.
ODI | Baseline and 3months
  ODI (Oxygen Desaturation Index) is the number of oxygen desaturation events per hour of sleep. The number of events per hour in which SpO₂ drops by a certain percentage, usually 3% or 4%. Usually it's zero times.
Nocturnal hypoxemia | Baseline and 3months
  Nocturnal hypoxemia is characterized by mean overnight oxygen saturation (mean SpO₂) during sleep, minimum oxygen saturation (minimum SpO₂) observed during sleep, percentage of time with SpO2<90%(% of total sleep time, %TST). We will investigate how much the SpO2 level decreases during a single sleep period and the duration of that decrease.
Arousals per hour (arousal index) | Baseline and 3months
  Arousals is an assessment of wakefulness events during sleep. The more times it occurs, the more it is thought to lead to a decline in sleep quality.
COPD assessment test: CAT | Baseline, 2months and 3months
  This questionnaire is designed for the simple assessment of symptoms and the impact on daily life in patients with COPD. It consists of eight items, each scored from 0 to 5. Higher scores indicate more severe symptoms and greater impact on daily life.
Hospital Anxiety and Depression Scale: HADS | Baseline, 2months and 3months
  The items are designed to be less influenced by physical symptoms, making them valid for patients with medical conditions. The total score for each is 0-21 points. A total score of 8 or more for odd numbers is considered a state of anxiety, and a total score of 11 or more for even numbers is considered a state of depression.
Number of technical errors | Baseline, 2months and 3 months
  For each inhalation device, the items in which the participant performs an incorrect inhalation technique are considered errors, and the number of such items is counted.

CONTACTS AND LOCATIONS:
Locations (1):
- Kumamoto University, Kumamoto, Chuo-ku, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moriyama M, Takeshita Y, Haruta Y, Hattori N, Ezenwaka CE. Effects of a 6-month nurse-led self-management program on comprehensive pulmonary rehabilitation for patients with COPD receiving home oxygen therapy. Rehabil Nurs. 2015 Jan-Feb;40(1):40-51. doi: 10.1002/rnj.119. Epub 2013 Aug 6. PMID 23922290
- [Result] Al-Kalaldeh M, El-Rahman MA, El-Ata A. Effectiveness of Nurse-Driven Inhaler Education on Inhaler Proficiency and Compliance Among Obstructive Lung Disease Patients: A Quasi-Experimental Study. Can J Nurs Res. 2016 Jun;48(2):48-55. doi: 10.1177/0844562116676119. PMID 28841042
- [Result] Sauriasari R, Madani RA, Rozaliyani A, Sudiana D. The effect of repeated education using live demonstrations and videos of how to use inhalation drugs on quality of life for COPD patients. Heliyon. 2021 Aug 24;7(9):e07870. doi: 10.1016/j.heliyon.2021.e07870. eCollection 2021 Sep. PMID 34504968
- [Result] Muller T, Muller A, Hubel C, Knipel V, Windisch W, Cornelissen CG, Dreher M. Optimizing inhalation technique using web-based videos in obstructive lung diseases. Respir Med. 2017 Aug;129:140-144. doi: 10.1016/j.rmed.2017.06.009. Epub 2017 Jun 17. PMID 28732821
- [Result] Ngo CQ, Phan DM, Vu GV, Dao PN, Phan PT, Chu HT, Nguyen LH, Vu GT, Ha GH, Tran TH, Tran BX, Latkin CA, Ho CSH, Ho RCM. Inhaler Technique and Adherence to Inhaled Medications among Patients with Acute Exacerbation of Chronic Obstructive Pulmonary Disease in Vietnam. Int J Environ Res Public Health. 2019 Jan 10;16(2):185. doi: 10.3390/ijerph16020185. PMID 30634631
- [Result] Ahn JH, Chung JH, Shin KC, Jin HJ, Jang JG, Lee MS, Lee KH. The effects of repeated inhaler device handling education in COPD patients: a prospective cohort study. Sci Rep. 2020 Nov 12;10(1):19676. doi: 10.1038/s41598-020-76961-y. PMID 33184428
- [Result] Lindh A, Theander K, Arne M, Lisspers K, Lundh L, Sandelowsky H, Stallberg B, Westerdahl E, Zakrisson AB. One additional educational session in inhaler use to patients with COPD in primary health care - A controlled clinical trial. Patient Educ Couns. 2022 Sep;105(9):2969-2975. doi: 10.1016/j.pec.2022.05.013. Epub 2022 May 26. PMID 35672192
- [Result] Bouloukaki I, Tzanakis N, Mermigkis C, Giannadaki K, Moniaki V, Mauroudi E, Michelakis S, Schiza SE. Tiotropium Respimat Soft Mist Inhaler versus HandiHaler to improve sleeping oxygen saturation and sleep quality in COPD. Sleep Breath. 2016 May;20(2):605-12. doi: 10.1007/s11325-015-1259-y. Epub 2015 Sep 25. PMID 26407963
- [Result] Krachman SL, Vega ME, Yu D, Demidovich J, Patel H, Jaffe F, Soler X, Shariff T, D'Alonzo GE, Chatila W, Weaver S, Daraz Y, Cohen S, Criner GJ. Effect of Triple Therapy with Budesonide-Formoterol-Tiotropium Versus Placebo-Tiotropium on Sleep Quality in Patients with Chronic Obstructive Pulmonary Disease. Chronic Obstr Pulm Dis. 2021 Apr 27;8(2):219-229. doi: 10.15326/jcopdf.2020.0178. PMID 33610139
- [Result] Sulaiman I, Seheult J, Sadasivuni N, MacHale E, Killane I, Giannoutsos S, Cushen B, Mokoka MC, Bhreathnach AS, Boland F, Reilly RB, Costello RW. The Impact of Common Inhaler Errors on Drug Delivery: Investigating Critical Errors with a Dry Powder Inhaler. J Aerosol Med Pulm Drug Deliv. 2017 Aug;30(4):247-255. doi: 10.1089/jamp.2016.1334. Epub 2017 Mar 9. PMID 28277810
- [Result] Lee SH, Kim KU, Lee H, Park HK, Kim YS, Lee MK. Sleep disturbance in patients with mild-moderate chronic obstructive pulmonary disease. Clin Respir J. 2019 Dec;13(12):751-757. doi: 10.1111/crj.13085. Epub 2019 Aug 30. PMID 31449723
- [Result] Czerwaty K, Dzaman K, Sobczyk KM, Sikorska KI. The Overlap Syndrome of Obstructive Sleep Apnea and Chronic Obstructive Pulmonary Disease: A Systematic Review. Biomedicines. 2022 Dec 21;11(1):16. doi: 10.3390/biomedicines11010016. PMID 36672523
- [Result] Azuma M, Chin K, Yoshimura C, Takegami M, Takahashi K, Sumi K, Nakamura T, Nakayama-Ashida Y, Minami I, Horita S, Oka Y, Oga T, Wakamura T, Fukuhara S, Mishima M, Kadotani H. Associations among chronic obstructive pulmonary disease and sleep-disordered breathing in an urban male working population in Japan. Respiration. 2014;88(3):234-43. doi: 10.1159/000366064. Epub 2014 Aug 22. PMID 25171691
- [Result] Climaco DCS, Lustosa TC, Silva MVFP, Lins-Filho OL, Rodrigues VK, Oliveira-Neto LAP, Feitosa ADM, Queiroga FJP Jr, Cabral MM, Pedrosa RP. Sleep quality in COPD patients: correlation with disease severity and health status. J Bras Pneumol. 2022 Apr 29;48(3):e20210340. doi: 10.36416/1806-3756/e20210340. eCollection 2022. PMID 35508063
- [Result] Lin L, Song Q, Duan J, Liu C, Cheng W, Zhou A, Peng Y, Zhou Z, Zeng Y, Chen Y, Cai S, Chen P. The impact of impaired sleep quality on symptom change and future exacerbation of chronic obstructive pulmonary disease. Respir Res. 2023 Mar 30;24(1):98. doi: 10.1186/s12931-023-02405-6. PMID 36998013
- [Result] Shorofsky M, Bourbeau J, Kimoff J, Jen R, Malhotra A, Ayas N, Tan WC, Aaron SD, Sin DD, Road J, Chapman KR, O'Donnell DE, Maltais F, Hernandez P, Walker BL, Marciniuk D, Kaminska M; Canadian Respiratory Research Network; CanCOLD Collaborative Research group. Impaired Sleep Quality in COPD Is Associated With Exacerbations: The CanCOLD Cohort Study. Chest. 2019 Nov;156(5):852-863. doi: 10.1016/j.chest.2019.04.132. Epub 2019 May 28. PMID 31150638
- [Result] Kwon JS, Wolfe LF, Lu BS, Kalhan R. Hyperinflation is associated with lower sleep efficiency in COPD with co-existent obstructive sleep apnea. COPD. 2009 Dec;6(6):441-5. doi: 10.3109/15412550903433000. PMID 19938967

DOCUMENTS (2):
  • Study Protocol (2025-06-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT07311499/Prot_000.pdf
  • Informed Consent Form (2025-06-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT07311499/ICF_001.pdf